CLINICAL TRIAL: NCT04704882
Title: A Modified Omental Patch Work Decreases Pancreatic Fistula After Laparoscopic Pancreaticoduodenectomy
Brief Title: A Modified Omental Patch Work Decreases Pancreatic Fistula After Lpd
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yi-Ping Mou, Professor, Zhejiang Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZJPPHGIP-RCT2019001
Record Dates: First submitted 2021-01-04; First posted 2021-01-12 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Omental Patch; Laparoscopic Pancreaticoduodenectomy; Pancreatic Fistula
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omental patchwork group (Experimental)
  Interventions: Other: omental patchwork
- non-omental patchwork group (No Intervention)

INTERVENTIONS:
Other: omental patchwork — the omental flaps were sewn to lesser omentum and hepatorenal ligament to cover all the vessels
  Arms: omental patchwork group

SUMMARY:
Pancreaticoduodenecotmy(PD) is considered as the standard procedure for peri-amplullary or pancreatic head tumors. Laparoscopic pancreaticoduodenctomy(LPD) has been reported with minimal invasive advantages, such as small incision, less blood loss, less pain, et al. Further, some trials showed LPD got less morbidity and shorter length of stay. Pancreatic fistula is the major complication for pancreaticodupdenectomy and associated with numerous serious complications, suffering reoperation or sometimes death. The reported rate was 10% to 55%. A lot of modified procedure have been proposed to reduce pancreatic fistula. Omental flaps around anastomosis have been used to prevent post pancreaticoduodenectomy fistula or hemorrhage. However, the outcomes are controversy. A modified omental patch work has been used during LPD and the initial outcomes are good. This is a pilot study to evaluate the function of the modified omental patch work on decreasing the pancreatic fistula.

ELIGIBILITY:
Inclusion Criteria:

1. . Disease of periampullary or pancreatic head tumor
2. . Age: 18 years or older
3. Distant metastases are not diagnosed preoperatively.
4. . Patients who can provide written informed consent

Exclusion Criteria:

1. . Patients with severe organ disease such as cardiac disease,respiratory illness
2. . Patients with extended LPD or vessels reconstruction
3. Patients with conversion to laparotomy
4. . Patients with pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
pancreatic fistula | 90 days
  Incidence of pancreatic fistula grade B/C defined by ISGPF classification

SECONDARY OUTCOMES:
morbidity | 90 days
Mortality | 90 days
Postoperative hospital stay | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People'S Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided